CLINICAL TRIAL: NCT03921528
Title: Phase 2 Active Treatment Study to Evaluate the Efficacy and Safety of SRK-015 in Patients With Later-Onset Spinal Muscular Atrophy (TOPAZ)
Brief Title: An Active Treatment Study of SRK-015 in Patients With Type 2 or Type 3 Spinal Muscular Atrophy
Acronym: TOPAZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scholar Rock, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRK-015-002
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Results first posted 2022-11-17 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Spinal Muscular Atrophy; Spinal Muscular Atrophy Type 3; Spinal Muscular Atrophy Type 2; SMA; Neuromuscular Diseases; Muscular Atrophy; Atrophy; Muscular Atrophy, Spinal; Neuromuscular Manifestations
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood; Neuromuscular Diseases; Muscular Atrophy; Atrophy; Neuromuscular Manifestations | interventions — apitegromab

STUDY DESIGN:
Masking Description: Active treatment, randomized, double-blind for Cohort 3
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Ambulatory Type 3 SMA
  Interventions: Biological: SRK-015
- Cohort 2 (Experimental): Type 2 SMA / Non-Ambulatory Type 3 SMA
  Interventions: Biological: SRK-015
- Cohort 3 (Experimental): Type 2 SMA
  Interventions: Biological: SRK-015

INTERVENTIONS:
Biological: SRK-015 — SRK-015 is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that binds to human pro/latent myostatin with high affinity. SRK-015 will be administered every 4 weeks by intravenous infusion.

SUMMARY:
The TOPAZ study will assess the safety and efficacy of SRK-015 in later-onset Spinal Muscular Atrophy (SMA Type 2 and Type 3) in pediatric and adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 through 21 years old at the time of screening for Cohorts 1 and 2; Age ≥2 years old at the time of screening for Cohort 3.
* Documented diagnosis of 5q SMA.
* Diagnosed as later-onset (e.g., Type 2 or Type 3) SMA prior to receiving any treatment with therapy approved for SMA.
* Non-ambulatory patients must be able to sit independently (sits up straight with head erect for at least 10 seconds; does not use arms or hands to balance body or support position) per World Health Organization (WHO) motor milestones definition at screening.
* Ambulatory patients must have the ability to independently ambulate without aids or orthotics over 10 meters in 30 seconds or less at screening.
* Receiving the same background SMA therapy (e.g., on an approved survival motor neuron (SMN) upregulator therapy such as nusinersen, or not on any SMA therapy) for at least 6 months prior to screening and anticipated to remain on that therapy throughout the duration of the study.

  * If receiving the SMN upregulator therapy nusinersen, must have completed the loading regimen and initiated maintenance dosing (i.e., completed at least one maintenance dose) with at least 4 weeks after the first maintenance dose having elapsed prior to screening.
* Nutritional status stable over the past 6 months and anticipated to be stable throughout the duration of the study.
* Have no physical limitations that would prevent the patient from undergoing motor function outcome measures throughout the duration of the study.
* Able to receive study drug infusions and provide blood samples through the use of a peripheral intravenous (IV) or a long-term IV access device that the patient has placed for reasons independent from the study throughout the duration of the study.
* Able to adhere to the requirements of the protocol, including travel to the study center and completing all study procedures and study visits.
* For patients who are expected to have reached reproductive maturity by the end of the study, adhere to study specific contraception requirements.

Exclusion Criteria:

* Use of tracheostomy with positive pressure.
* Use of chronic daytime non-invasive ventilatory support for >16 hours daily in the 2 weeks prior to dosing, or anticipated to regularly receive such daytime ventilator support chronically over the duration of the study.
* Any acute or co-morbid condition interfering with the well-being of the patient within 14 days of screening, including active systemic infection, the need for acute treatment or inpatient observation due to any reason.
* Severe scoliosis and/or contractures at screening. Based on clinical judgement, any scoliosis or contractures present must be stable over the past 6 months, anticipated to be stable for the duration of the study and not prevent the patient from being evaluated on any functional outcome measures throughout the duration of the study.
* Pregnant or breastfeeding.
* Major orthopedic or other interventional procedure, including spine or hip surgery, considered to have the potential to substantially limit the ability of the patient to be evaluated on any functional outcome measures, within 6 months prior to screening, or anticipated for the duration of the study.
* Prior history of a hypersensitivity reaction to a monoclonal antibody (mAb) or recombinant protein bearing an Fc domain (such as a soluble receptor- Fc fusion protein).
* Use of systemic corticosteroids within 60 days prior to screening. Inhaled or topical steroids are allowed.
* Treatment with investigational drugs within 3 months prior to screening.
* Use of therapies with potentially significant muscle effects (such as androgens, insulin-like growth factor, growth hormone, systemic betaagonist, botulinum toxin, or muscle relaxants) or muscle-enhancing supplements within 60 days prior to screening.
* Patient has any other condition, which in the opinion of the Investigator may compromise safety or compliance, would preclude the patient from successful completion of the study, or interfere with the interpretation of the results.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O. Crawford, MD, Principal Investigator — Johns Hopkins University
Locations (16):
- United States (11):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - The Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Columbia University, New York, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Childrens Medical Center Dallas, Dallas, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
- Italy (2):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Centro Clinico Nemo Pediatrico Policlinico A. Gemelli-Università Cattolica Sacro Cuore, Roma
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Spain (2):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crawford TO, Darras BT, Day JW, Dunaway Young S, Duong T, Nelson LL, Barrett D, Song G, Bilic S, Cote S, Sadanowicz M, Iarrobino R, Xu TJ, O'Neil J, Rossello J, Place A, Kertesz N, Nomikos G, Chyung Y. Safety and Efficacy of Apitegromab in Patients With Spinal Muscular Atrophy Types 2 and 3: The Phase 2 TOPAZ Study. Neurology. 2024 Mar 12;102(5):e209151. doi: 10.1212/WNL.0000000000209151. Epub 2024 Feb 8. PMID 38330285

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Monotherapy: Ambulatory Type 3 SMA apitegromab (SRK-015) 20mg/kg
  SRK-015: SRK-015 is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that binds to human pro/latent myostatin with high affinity. SRK-015 was administered every 4 weeks by intravenous infusion.
- Cohort 1 - Dual Therapy: Ambulatory Type 3 SMA apitegromab (SRK-015) + nusinersen
  SRK-015: SRK-015 is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that binds to human pro/latent myostatin with high affinity. SRK-015 was administered every 4 weeks by intravenous infusion.
- Cohort 2: Type 2 SMA / Non-Ambulatory Type 3 SMA apitegromab (SRK-015) 20 mg/kg + nusinersen
  SRK-015: SRK-015 is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that binds to human pro/latent myostatin with high affinity. SRK-015 was administered every 4 weeks by intravenous infusion.
- Cohort 3 - Low Dose: Type 2 SMA apitegromab (SRK-015) 2 mg/kg + nusinersen
  SRK-015: SRK-015 is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that binds to human pro/latent myostatin with high affinity. SRK-015 was administered every 4 weeks by intravenous infusion.
- Cohort 3 - High Dose: Type 2 SMA apitegromab (SRK-015) 20mg/kg + nusinersen
  SRK-015: SRK-015 is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that binds to human pro/latent myostatin with high affinity. SRK-015 was administered every 4 weeks by intravenous infusion.
Period: Overall Study
Arm/Group | Cohort 1 - Monotherapy | Cohort 1 - Dual Therapy | Cohort 2 | Cohort 3 - Low Dose | Cohort 3 - High Dose
Started | 11 | 12 | 15 | 10 | 10
Completed | 6 | 10 | 13 | 10 | 10
Not Completed | 5 | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Set: All participants who were enrolled/randomized and received at least 1 dose of study drug.
Groups:
- Cohort 1 - Dual Therapy: Ambulatory Type 3 SMA apitegromab (SRK-015) 20mg/kg + nusinersen
  SRK-015: SRK-015 is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that binds to human pro/latent myostatin with high affinity. SRK-015 was administered every 4 weeks by intravenous infusion.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Monotherapy | Cohort 1 - Dual Therapy | Cohort 2 | Cohort 3 - Low Dose | Cohort 3 - High Dose | Total
Number analyzed (Participants) | 11 | 12 | 15 | 10 | 10 | 58
Age, Continuous [Mean (Full Range); unit: Years] | 12.1 [7 to 19] | 13.1 [7 to 21] | 11.7 [8 to 19] | 4.1 [2 to 6] | 3.8 [2 to 6] | 9.67 [2 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 8 | 3 | 5 | 31
  Male | 3 | 5 | 7 | 7 | 5 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 0 | 1 | 5
  Not Hispanic or Latino | 11 | 10 | 13 | 10 | 9 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 0 | 2 | 0 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 2
  White | 5 | 12 | 12 | 10 | 8 | 47
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Change From Baseline in the Revised Hammersmith Scale (RHS) Total Score at Day 364 (Visit 15) [Month 12]
Description: The Revised Hammersmith Scale (RHS) is a 36 item clinical assessment of physical abilities in patients with Type 2 SMA and ambulatory or nonambulatory patients with Type 3 SMA. For the ambulatory Type 3 patients 5-21 years of age in Cohort 1 (N=23), the primary endpoint was the change from baseline in RHS total score at month 12. The RHS has a minimum achievable score of 0 and a maximum achievable score of 69. The RHS includes 33 items that are graded on a scale of 0, 1, 2, where 0 denotes the lowest level and 2 denotes the highest level of ability/function. The remaining 3 items are scored 0 or 1, where 0 denotes an inability and 1 denotes an ability to achieve. Higher scores indicate increased motor function. A positive change from Baseline indicates improvement.
Time Frame: Baseline up to 12 months
Population: The ITT Population: all enrolled/randomized patients who receive at least 1 dose of study drug. The ITT Population was the main population for analysis of efficacy endpoints; the analysis includes all assessments from all patients with the exception of assessments after missing 3 consecutive doses due to site access restrictions caused by COVID-19. The last observation carried forward (LOCF) method was used to impute the 12-month primary endpoint for data missing for other reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 - Monotherapy | Cohort 1 - Dual Therapy
Number analyzed (Participants) | 11 | 12
score on a scale | -0.1 (5.01) | 0.0 (2.56)

2. Primary Outcome: Cohort 2 and Cohort 3: Change From Baseline in Hammersmith Functional Motor Scale Expanded (HFMSE) Total Score at Day 364 (Visit 15) [Month 12]
Description: Cohort 2: For the nonambulatory Type 2 and Type 3 patients 5-21 years of age in Cohort 2 (N=15), the primary efficacy endpoint was the change from baseline in HFMSE total score at month 12.
  Cohort 3: For the nonambulatory Type 2 patients ≥2 years of age in Cohort 3 (N=20), the primary efficacy endpoint was the change from baseline in HFMSE total score at month 12.
  The Hammersmith Functional Motor Scale Expanded (HFMSE) assesses the physical abilities of patients with Type 2 and Type 3 SMA comprises 33 items graded on a scale of 0, 1, or 2, where 0 denotes unable, 1 denotes performed with modification or adaptation, and 2 denotes performed without modification or adaptation.
Time Frame: Baseline up to 12 months
Population: The ITT Population: all enrolled/randomized patients who receive at least one dose of study drug. The ITT Population was the main population for analysis of efficacy endpoints; the analysis included all assessments from all patients with the exception of assessments after missing 3 consecutive doses due to site access restrictions caused by COVID-19. The last observation carried forward (LOCF) method was used to impute the 12-month primary endpoint for data missing for other reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 2 | Cohort 3 - Low Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 14 | 9 | 8
score on a scale | 0.6 (3.5) | 5.3 (8.93) | 7.1 (6.42)

3. Secondary Outcome: Cohort 1:Change From Baseline in the Revised Hammersmith Scale (RHS) Total Score at Other Prespecified Timepoints
Description: The Revised Hammersmith Scale (RHS) is a 36 item clinical assessment of physical abilities in patients with Type 2 SMA and ambulatory or nonambulatory patients with Type 3 SMA; it has a maximum achievable score of 69. The RHS includes 33 items that are graded on a scale of 0, 1, 2, where 0 denotes the lowest level and 2 denotes the highest level of ability/function. The remaining 3 items are scored 0 or 1, where 0 denotes an inability and 1 denotes an ability to achieve.
Time Frame: Baseline to 12 months
Population: 1 patient in Cohort 1 Monotherapy did not complete Physical Therapy Assessments at V6 due to site imposed COVID-19 restrictions.
  1 patient in Cohort 1 Dual Therapy withdrew consent following discontinuation of apitegromab after 3 months of treatment due to a nonserious TEAE of unresolved fatigue assessed as not related to apitegromab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Monotherapy | Cohort 1 - Dual Therapy
Number analyzed (Participants) | 11 | 12
Participants
  ≥5pt at Day 56 (V4) | 1 | 1
  ≥5pt at Day 112 (V6): number analyzed (Participants) | 10 | 11
  ≥5pt at Day 112 (V6) | 1 | 1
  ≥5pt at Day 168 (V8): number analyzed (Participants) | 11 | 11
  ≥5pt at Day 168 (V8) | 2 | 1
  ≥5pt Month 12 Endpoint | 1 | 0
  ≥3pt at Day 56 (V4) | 3 | 3
  ≥3pt at Day 112 (V6): number analyzed (Participants) | 10 | 11
  ≥3pt at Day 112 (V6) | 1 | 2
  ≥3pt at Day 168 (V8): number analyzed (Participants) | 11 | 11
  ≥3pt at Day 168 (V8) | 4 | 1
  ≥3pt at Month 12 Endpoint | 3 | 3
  ≥1pt at Day 56 (V4) | 8 | 8
  ≥1pt at Day 112 (V6): number analyzed (Participants) | 10 | 11
  ≥1pt at Day 112 (V6) | 3 | 5
  ≥1pt at Day 168 (V8): number analyzed (Participants) | 11 | 11
  ≥1pt at Day 168 (V8) | 7 | 4
  ≥1pt at Month 12 Endpoint | 6 | 5
  No Change at Day 56 (V4) | 1 | 1
  No Change at Day 112 (V6): number analyzed (Participants) | 10 | 11
  No Change at Day 112 (V6) | 5 | 1
  No Change at Day 168 (V8): number analyzed (Participants) | 11 | 11
  No Change at Day 168 (V8) | 1 | 5
  No Change at Month 12 Endpoint | 0 | 2
  Decrease at Day 56 (V4) | 2 | 3
  Decrease at Day 112 (V6): number analyzed (Participants) | 10 | 11
  Decrease at Day 112 (V6) | 2 | 5
  Decrease at Day 168 (V8): number analyzed (Participants) | 11 | 11
  Decrease at Day 168 (V8) | 3 | 2
  Decrease at Month 12 Endpoint | 5 | 5

4. Secondary Outcome: Cohort 1: Proportion of Patients Achieving Various Magnitudes of Change in RHS Score From Baseline
Description: as for outcome 3
Time Frame: Baseline to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Monotherapy | Cohort 1 - Dual Therapy
Number analyzed (Participants) | 11 | 12
Participants
  ≥3pt increase | 3 | 3
  ≥1pt increase | 6 | 5
  No Change | 0 | 2
  Decrease | 5 | 5

5. Secondary Outcome: Cohort 1: Change From Baseline in 6-Minute Walk Test (6MWT)
Description: 6-Minute Walk Test The 6-Minute Walk Test (6MWT) is an assessment of exercise capacity and fatigue used for ambulatory patients with later-onset SMA who are directed to walk along a 25 meter course as fast as possible over 6 minutes.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Cohort 1 - Monotherapy | Cohort 1 - Dual Therapy
Number analyzed (Participants) | 8 | 11
Meters | -20.6 (44.96) | 11.0 (33.67)

6. Secondary Outcome: Cohort 1: Change From Baseline in 30-Second Sit-to-Stand
Description: The 30-Second Sit-to-Stand Test is an assessment of functional lower-limb strength that measures the maximal number of times a patient can transition from sitting to standing in 30 seconds.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: Stands
Arm/Group | Cohort 1 - Monotherapy | Cohort 1 - Dual Therapy
Number analyzed (Participants) | 11 | 12
Stands | -0.6 (1.63) | -0.2 (1.95)

7. Secondary Outcome: Cohort 1: Change From Baseline in 10-Meter Walk/Run (From RHS)
Description: The 10 Meter Walk/Run test is an enhanced function of the RHS used for ambulatory patients with Type 3 SMA. It is a measure of the time taken to walk/run 10 meters. The time to perform is summarized only for patients able to complete the RHS 10-meter walk/run item.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort 1 - Monotherapy | Cohort 1 - Dual Therapy
Number analyzed (Participants) | 7 | 11
Seconds | 0.1 (0.32) | 0.9 (3.32)

8. Secondary Outcome: Cohort 1: Change From Baseline in Timed Rise From Floor (From RHS)
Description: The timed rise from floor test is an enhanced function of the RHS used for ambulatory patients with Type 3 SMA. It is a measure of the time taken to rise to standing from the floor. The time to rise from floor is summarized only for patients able to complete the RHS rise from floor item.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cohort 1 - Monotherapy | Cohort 1 - Dual Therapy
Number analyzed (Participants) | 5 | 6
Seconds | 0.6 (1.75) | -0.6 (1.43)

9. Secondary Outcome: Cohort 2 &3: Change From Baseline in HFMSE Total Score at Other Prespecified Timepoints
Description: The Hammersmith Functional Motor Scale Expanded (HFMSE) assesses the physical abilities of patients with Type 2 and Type 3 SMA comprises 33 items graded on a scale of 0, 1, or 2, where 0 denotes unable, 1 denotes performed with modification or adaptation, and 2 denotes performed without modification or adaptation.
Time Frame: Baseline to 12 months
Population: 1 patient in Cohort 2 and 3 patients in Cohort 3 (1 low dose and 2 high dose) missed 3 consecutive doses of apitegromab during the 12-month treatment period due to COVID-19-related site access restrictions and were not included in the primary analysis. In addition, 2 cohort 3 low dose patients skipped motor assessments at Day 168 (V8) and 1 cohort low dose patient at Day 365 (V15) due to COVID restrictions.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 | Cohort 3 - Low Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 15 | 10 | 10
Participants
  ≥5pt at Day 56 (V4) | 1 | 0 | 3
  ≥5pt at Day 112 (V6): number analyzed (Participants) | 14 | 10 | 10
  ≥5pt at Day 112 (V6) | 1 | 2 | 5
  ≥5pt at Day 168 (V8): number analyzed (Participants) | 14 | 7 | 8
  ≥5pt at Day 168 (V8) | 1 | 3 | 4
  ≥5pt at Month 12 Endpoint: number analyzed (Participants) | 14 | 9 | 8
  ≥5pt at Month 12 Endpoint | 2 | 5 | 5
  ≥3pt at Day 56 (V4) | 1 | 4 | 5
  ≥3pt at Day 112 (V6): number analyzed (Participants) | 14 | 10 | 10
  ≥3pt at Day 112 (V6) | 2 | 3 | 5
  ≥3pt at Day 168 (V8): number analyzed (Participants) | 14 | 7 | 8
  ≥3pt at Day 168 (V8) | 2 | 4 | 5
  ≥3pt at Month 12 Endpoint: number analyzed (Participants) | 14 | 9 | 8
  ≥3pt at Month 12 Endpoint | 4 | 5 | 5
  ≥1pt at Day 56 (V4) | 4 | 6 | 8
  ≥1pt at Day 112 (V6): number analyzed (Participants) | 14 | 10 | 10
  ≥1pt at Day 112 (V6) | 6 | 5 | 9
  ≥1pt at Day 168 (V8): number analyzed (Participants) | 14 | 7 | 8
  ≥1pt at Day 168 (V8) | 10 | 5 | 8
  ≥1pt at Month 12 Endpoint: number analyzed (Participants) | 14 | 9 | 8
  ≥1pt at Month 12 Endpoint | 9 | 7 | 7
  No Change at Day 56 (V4) | 4 | 1 | 1
  No Change at Day 112 (V6): number analyzed (Participants) | 14 | 10 | 10
  No Change at Day 112 (V6) | 5 | 2 | 1
  No Change at Day 168 (V8): number analyzed (Participants) | 14 | 7 | 8
  No Change at Day 168 (V8) | 1 | 1 | 0
  No Change at Month 12 Endpoint: number analyzed (Participants) | 14 | 9 | 8
  No Change at Month 12 Endpoint | 1 | 0 | 0
  Decrease at Day 56 (V4) | 7 | 3 | 1
  Decrease at Day 112 (V6): number analyzed (Participants) | 14 | 10 | 10
  Decrease at Day 112 (V6) | 3 | 3 | 0
  Decrease at Day 168 (V8): number analyzed (Participants) | 14 | 7 | 8
  Decrease at Day 168 (V8) | 3 | 1 | 0
  Decrease at Month 12 Endpoint: number analyzed (Participants) | 14 | 9 | 8
  Decrease at Month 12 Endpoint | 4 | 2 | 1

10. Secondary Outcome: Cohort 2 & 3: Proportion of Patients Achieving Various Magnitudes of Change in HFMSE Score From Baseline
Description: as for outcome 9
Time Frame: Baseline to 12 months
Population: 1 patient in Cohort 2 and 3 patients in Cohort 3 missed 3 consecutive doses of apitegromab during the 12-month treatment period due to COVID-19-related site access restrictions and were not included in the primary analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 | Cohort 3 - Low Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 14 | 9 | 8
Participants
  ≥3pt increase | 4 | 5 | 5
  ≥1pt increase | 9 | 7 | 7
  No Change | 1 | 0 | 0
  Decrease | 4 | 2 | 1

11. Secondary Outcome: Cohort 2 & 3: Change in Baseline in Revised Upper Limb Module (RULM) Total Score
Description: The RULM is a 20 item assessment of upper limb function in nonambulatory patients with SMA that was performed for patients who were 30 months of age or older at baseline. The 19 scored items assess functions that relate to everyday life, such as pressing a button and picking up a token; these items are scored 0, 1, or 2, where 0 denotes unable, 1 denotes able with modification, and 2 denotes able with no modification. The maximum score achievable is 37.
Time Frame: Baseline to 12 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Cohort 2 | Cohort 3 - Low Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 14 | 9 | 8
Score on scale | 1.2 (2.99) | 0.9 (2.62) | 1 (2.94)

12. Secondary Outcome: Cohort 2 & 3: Proportion of Patients Achieving a New WHO Motor Development Milestones Relative to Baseline
Description: The WHO Multicenter Growth Reference Study performance criteria is being utilized to assess the World Health Organization (WHO) motor development milestones of patients with Type 2 and nonambulatory Type 3 SMA enrolled in Cohort 2 and Cohort 3 relative to baseline. The WHO milestone assessment consists of six items which were selected because they have been considered to be universal, fundamental, and simple to test and evaluate, they include 1) sitting without support, 2) hands and knees crawling, 3) standing with assistance, 4) walking with assistance, 5) standing alone, and 6) walking without assistance. Each item is recorded as 1 (unable), 2 (refusal), 3 (Yes) or 9 (did not test). The number of 3s was counted as the final score. The minimum was 0, which means no motor milestones were achieved; the maximum was 6, which means all 6 milestones were achieved.
Time Frame: Baseline to 12 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 | Cohort 3 - Low Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 14 | 9 | 8
Participants
  ≥2pt increase | 1 | 0 | 1
  ≥1pt increase | 3 | 1 | 1
  No Change | 11 | 7 | 6
  Decrease | 0 | 1 | 1

13. Secondary Outcome: Cohort 2 & 3: Proportion of Patients Achieving Various Magnitudes of Change in RULM Score From Baseline
Description: as for outcome 11
Time Frame: Baseline to 12 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 | Cohort 3 - Low Dose | Cohort 3 - High Dose
Number analyzed (Participants) | 14 | 9 | 7
Participants
  ≥2pt increase | 5 | 3 | 2
  ≥1pt increase | 8 | 3 | 3
  No change | 1 | 3 | 2
  Decrease | 5 | 3 | 2

ADVERSE EVENTS:
Time Frame: Day 0 (Visit 1) to 48 months (Visit EC14)
Description: Classification based on the FDA regulatory definition of an AE.
Groups:
- Cohort 1 - Monotherapy: Ambulatory Type 3 SMA apitegromab (SRK-015) 20 mg/kg
  SRK-015: SRK-015 is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that binds to human pro/latent myostatin with high affinity. SRK-015 was administered every 4 weeks by intravenous infusion.
- Cohort 1 - Dual Therapy: Ambulatory Type 3 SMA apitegromab (SRK-015) 20 mg/kg + nusinersen
  SRK-015: SRK-015 is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that binds to human pro/latent myostatin with high affinity. SRK-015 was administered every 4 weeks by intravenous infusion.
- Cohort 2: Type 2 SMA / Non-Ambulatory Type 3 SMA apitegromab (SRK-015) 20mg/kg + nusinersen
  SRK-015: SRK-015 is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that binds to human pro/latent myostatin with high affinity. SRK-015 was administered every 4 weeks by intravenous infusion.
- Cohort 3 - High Dose: Type 2 SMA apitegromab (SRK-015) 20 mg/kg + nusinersen
  SRK-015: SRK-015 is a fully human anti-proMyostatin monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/lambda isotype that binds to human pro/latent myostatin with high affinity. SRK-015 was administered every 4 weeks by intravenous infusion.
Arm/Group | Cohort 1 - Monotherapy | Cohort 1 - Dual Therapy | Cohort 2 | Cohort 3 - Low Dose | Cohort 3 - High Dose
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/15 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 4/11 | 4/12 | 9/15 | 6/10 | 5/10
Other Adverse Events (participants affected / at risk) | 11/11 | 11/12 | 15/15 | 10/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Monotherapy (N=11) | Cohort 1 - Dual Therapy (N=12) | Cohort 2 (N=15) | Cohort 3 - Low Dose (N=10) | Cohort 3 - High Dose (N=10)
Gait Inability (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post Lumbar-Puncture Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenoidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hospitalization (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation reduction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Scoliosis surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 1 (1)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Monotherapy (N=11) | Cohort 1 - Dual Therapy (N=12) | Cohort 2 (N=15) | Cohort 3 - Low Dose (N=10) | Cohort 3 - High Dose (N=10)
Upper respiratory tract infection (Infections and infestations) | 5 (9) | 5 (9) | 5 (10) | 4 (12) | 5 (10)
Nasopharyngitis (Infections and infestations) | 4 (5) | 1 (5) | 6 (13) | 6 (23) | 5 (19)
Influenza (Infections and infestations) | 3 (4) | 1 (1) | 3 (3) | 3 (5) | 3 (3)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (9) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 5 (5) | 6 (10) | 4 (18) | 9 (37)
Fatigue (General disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 1 (2) | 2 (6) | 6 (11) | 8 (21)
Nausea (Gastrointestinal disorders) | 4 (8) | 3 (4) | 3 (4) | 5 (7) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 0 (0) | 3 (4) | 2 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (4) | 2 (6) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5) | 4 (5) | 5 (18) | 7 (22)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (6) | 2 (3) | 2 (5) | 4 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 3 (10) | 4 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 3 (4) | 2 (4) | 4 (12)
Scoliosis (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4) | 5 (6) | 1 (1) | 3 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (5) | 3 (4) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (8) | 1 (1) | 3 (4) | 0 (0) | 2 (5)
Headache (Nervous system disorders) | 7 (10) | 5 (14) | 5 (18) | 4 (8) | 3 (9)
Dizziness (Nervous system disorders) | 4 (10) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1) | 4 (5) | 3 (3) | 4 (9)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (11) | 6 (54) | 1 (1) | 2 (3) | 1 (2)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 3 (5) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gait Inability (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Administration site conditions
Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (3) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Astigmatism (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excessive eye blinking (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eyelid disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (4) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Gingival ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site rash (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — General disorders and administration site conditions
Asthenia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — General disorders and administration site conditions
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait inability (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperpyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infusion site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tissue infiltration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vessel puncture site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site injury (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Injection site pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 3 (4) | 6 (7) | 6 (7) | 6 (6)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis genital (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heliobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Norovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (4) | 1 (1) | 2 (2) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Rhinitis (Infections and infestations) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Animal scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthopod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood ketone body (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone density decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calcium deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Feeding disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 5 (11) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 4 (4)
Hip deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint laxity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuromuscular scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain fog (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autism spectrum disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autism spectrum disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fear of injection (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypohidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rash follicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin striae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle operation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 45 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT03921528/Prot_SAP_000.pdf